CLINICAL TRIAL: NCT00262197
Title: Patient Based Strategy to Reduce Errors in Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 0105300; U18HS011919 (AHRQ)
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Medical error rates; Pharmacotherapy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Customized Physician Intervention
Behavioral: Customized Patient Intervention

SUMMARY:
This project evaluates a HPMG effort to reduce error rates through customized direct feedback of diabetes quality of care data to diabetes patients and their physicians. HPMG has routinely provided patients with personalized feedback of glucose and cholesterol test results since about 1997. This project will implement and evaluate the impact of this intervention on diabetes medical error rates and resource use.

DETAILED DESCRIPTION:
The project, Patient-Based Strategy to Reduce Errors in Diabetes Care (referred to as MOVES), addresses issues of overuse, under use, or misuse of care for adults with diabetes. This combination research and translation project has been developed as a component of the Pursuing Perfection initiative of HealthPartners Medical Group, with the close collaboration of HPMG leadership. HealthPartners Medical Group is widely regarded as a national leader in diabetes care, with dramatic improvements in both glucose control and cholesterol control over the past 8 years [Graphs].

The MOVES study is attempting to activate patients with diabetes to be more involved in their care. To help patients do this, HPMG sends patients a customized summary of their care. The summary includes a graph of recent glucose and cholesterol test results and specific suggestions that may improve care. In many cases, a visit with the patient's personal physician is encouraged to assure ongoing progress towards important evidence-based goals in diabetes care.

Physicians also receive a matched communication that indicates areas for potential improvement and makes technical suggestions for care based on the Staged Diabetes Management © protocols. The project tries to ally expert judgment with the physician's personal knowledge of a patient. It is felt that this approach is critical to assessing what the best improvement strategy may be in each individual case.

This inexpensive customized intervention has potential to be widely disseminated and can be seamlessly integrated with other interventions to further achievement of clinical goals. The results are relevant to patients, clinicians, payers, and policymakers.

ELIGIBILITY:
Inclusion Criteria:

* For physician intervention inclusion criteria included; 1)primary care (general internist or family) physician in HealthPartners Medical Group. 2)Provided ongoing care to 20 or more adult patients with diabetes.
* For patients inclusion criteria included; An established diagnosis of diabetes based on either (a) two or more ICD-9 diagnosis codes for diabetes in a 12-month period of time, or (b) a filled prescription for a diabetes-specific drug within a 12-month period of time.

In addition, participating patients met all of the following criteria: (a) age less than 75 years, (b) Charlson comorbidity score of 3 or less, (c) linked to the a primary care physician who was participating in the study in two consecutive calendar years, (d) had pharmacy coverage at the time of the intervention and for the previous 12-month period, and (e) had either HBA1c > 7% or LDL > 130 mg/dl (or LDL > 100 mg/dl if the patient also had CHD).

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000
Dates: Start 2001-12; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The following dependant variables were measured in this study;
Diabetes medical error in the 12 months post-intervention, Glycated hemoglobin (A1c) values and A1c test rates in the 12 months post-intervention, and
LDL-cholesterol levels and test rates in the 12 months post-intervention.

SECONDARY OUTCOMES:
Age
Gender
Charlson comorbidity score

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, MD, MPH, Principal Investigator — HealthPartners Institute

REFERENCES:
- [Background] Sperl-Hillen JM, O'Connor PJ. Factors driving diabetes care improvement in a large medical group: ten years of progress. Am J Manag Care. 2005 Aug;11(5 Suppl):S177-85. PMID 16111440
- [Background] O'Connor PJ, Gray RJ, Maciosek MV, Fillbrandt KM, DeFor TA, Alexander CM, Weiss TW, Teutsch SM. Cholesterol levels and statin use in patients with coronary heart disease treated in primary care settings. Prev Chronic Dis. 2005 Jul;2(3):A05. Epub 2005 Jun 15. PMID 15963307
- [Background] Gilmer TP, O'Connor PJ, Rush WA, Crain AL, Whitebird RR, Hanson AM, Solberg LI. Predictors of health care costs in adults with diabetes. Diabetes Care. 2005 Jan;28(1):59-64. doi: 10.2337/diacare.28.1.59. PMID 15616234
- [Background] O'Connor PJ, Sperl-Hillen JM, Johnson PE, Rush WA, Biltz G. Clinical Inertia and Outpatient Medical Errors. In: Henriksen K, Battles JB, Marks ES, Lewin DI, editors. Advances in Patient Safety: From Research to Implementation (Volume 2: Concepts and Methodology). Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK20513/ PMID 21249838
- [Background] O'Connor PJ, Sperl-Hillen JM, Johnson PE, Rush WA. Identification, Classification, and Frequency of Medical Errors in Outpatient Diabetes Care. In: Henriksen K, Battles JB, Marks ES, Lewin DI, editors. Advances in Patient Safety: From Research to Implementation (Volume 1: Research Findings). Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK20464/ PMID 21249801
- [Derived] O'Connor PJ, Sperl-Hillen J, Johnson PE, Rush WA, Crain AL. Customized feedback to patients and providers failed to improve safety or quality of diabetes care: a randomized trial. Diabetes Care. 2009 Jul;32(7):1158-63. doi: 10.2337/dc08-2247. Epub 2009 Apr 14. PMID 19366977